CLINICAL TRIAL: NCT02455596
Title: Phase II Study of Recombinant Anti-tumor and Anti-virus Protein for Injection to Treat Advanced Neuroendocrine Tumors
Brief Title: Recombinant Anti-tumor and Anti-virus Protein for Injection to Treat Advanced Neuroendocrine Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JH-NETs-001
Record Dates: First submitted 2015-05-21; First posted 2015-05-28 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2015-10

CONDITIONS: Neuroendocrine Tumors
Keywords: Novaferon; Recombinant anti-tumor and anti-virus protein for injection; Carcinoid Tumor; Pancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Adenoma, Islet Cell | interventions — Injections; recombinant interferon alpha 2b-like protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Recombinant anti-tumor and anti-virus protein for injection(Novaferon), three times per week.
  Interventions: Drug: Recombinant anti-tumor and anti-virus protein for injection (Novaferon)

INTERVENTIONS:
Drug: Recombinant anti-tumor and anti-virus protein for injection (Novaferon) — Recombinant anti-tumor and anti-virus protein for injection, 10μg, im, 3 times for first week,followed by 20μg for two weeks, and followed a maintenance dose of 30μg, the frequency of administration is three times per week.
  Other Names: Novaferon

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of recombinant anti-tumor and anti-virus protein for injection in treating patients with advanced neuroendocrine tumors who have failed standard treatment or are unable to receive standard treatment.

DETAILED DESCRIPTION:
This is a Phase Ⅱ exploratory clinical study. The purpose of this study is to evaluate the efficacy and safety of recombinant anti-tumor and anti-virus protein for injection in treating patients with advanced neuroendocrine tumors who have failed standard treatment or are unable to receive standard treatment.

Recombinant anti-tumor and anti-virus protein for injection, 10μg,im,3 times for the first week, followed by 20μg for two weeks, and followed a maintenance dose of 30μg, the frequency of administration is three times per week. Treatment continued until the patient died or had unacceptable toxicity or had disease progression or required to discontinue the treatment. At the time of disease progression, if investigators believe patients can continue to benefit from the investigational product, patients may be provided with recombinant anti-tumor and anti-virus protein for injection,but only survival follow-up datas will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Have been fully aware of the study and voluntarily signed the informed consent.
* At least 18 years old.
* Have a confirmed histological or cytological diagnosis of low- or intermediate-grade advanced NETs (unresectable or metastatic), the pathology must meet one of the following criteria: (a) primary site of lung or thymus (carcinoid) with mitotic count of ≤ 10/10 High Power Field [HPF]) (b) other primary site (including primary unknown) with mitotic count of ≤ 20/10 High Power Field [HPF] and Ki67 index of ≤ 20%，or with Ki67 index of > 20% and well-differentiated.
* Patients who have failed standard treatment or are unable to receive standard treatment, and have disease progression within the past 12 months;
* At least one measurable lesion according to the RECIST 1.1 criteria that has not been previously locally treated.
* ECOG performance status 0, 1 or 2.
* Minimum of 4 weeks since any local radiotherapy or surgery for the control of symptoms or severe complications(local radiotherapy for the control of bone metastases is not the limit)，and adequately recovered from toxicities of any prior therapy).
* Life expectancy of at least 3 months.

Exclusion Criteria:

* Prior treatment with Recombinant Anti-tumor and Anti-virus Protein for Injection.
* Prior treatment with Interferon.
* Pregnancy or breast-feeding women or women who may be pregnant were positive drug test before administration.
* Patient of child-bearing potential(male or less than 1 year postmenopausal women) were reluctant to take contraceptive measures.
* Patient who were allergic to Interferon-α or who had interferon-α antibody.
* Have brain metastases or previous history of brain metastases or history of seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1 year
  PFS is defined as the length of time from random assignment to disease progression or to death resulting from any cause other than the progress.
Disease control rate(DCR) | 1 year
  DCR is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response + Stable Disease as best overall response according to radiological assessments.

SECONDARY OUTCOMES:
Overall response rate(ORR) | 1 year
  ORR is defined as the percentage of subjects having achieved confirmed Complete Response + Partial Response as best overall response according to radiological assessments.
Overall survival (OS) | 3 years
  OS is defined as the length of time from random assignment to death or to last contact
Adverse Events(AEs) | 1 year
  AEs are evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Jianming, M.D., Principal Investigator — 307 Hospital of PLA
Locations (1):
- 307 Hospital of PLA, Beijing, Beijing Municipality, China